CLINICAL TRIAL: NCT02941653
Title: Effect of Potassium Oxalate and Potassium Nitrate on Tooth Sensitivity Related to in Office Bleaching: Randomized Clinical Trial
Brief Title: Potassium Oxalate and Potassium Nitrate and Post-bleaching Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, Flavia Pardo Salata Nahsan, Principal Investigator, Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFSergipeHU
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Medicaments Substances in Therapeutic Use

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control: Potassium Nitrate 2% gel (Active Comparator): The patient will receive the application of potassium nitrate 2% gel on vestibular surface teeth, for 10 minutes.
  Interventions: Device: Potassium nitrate 2% gel
- Intervention: Potassium Oxalate 5% gel (Experimental): The patient will receive the application of potassium oxalate 5% gel on vestibular surface teeth, for 10 minutes.
  Interventions: Device: Potassium oxalate 5% gel

INTERVENTIONS:
Device: Potassium nitrate 2% gel — * Teeth will be cleaned using rubber cups associated to pumice and water;
  * Relative isolation with roller cotton will be done;
  * Prior to each bleaching session, the patients will receive the potassium nitrate 2% desensitivity gel application on vestibular surface, for 10 minutes.
  * Gingival dam will be performed using a fluid resin (Top Dam, FGM, Brazil)
  * A 35% hydrogen peroxide based bleaching agent will be mixed and applied on the vestibular surface of teeth, remaining for 40 minutes.
  Arms: Control: Potassium Nitrate 2% gel
Device: Potassium oxalate 5% gel — * Teeth will be cleaned using rubber cups associated to pumice and water
  * Relative isolation with roller cotton will be done;
  * Prior to each bleaching session, the patients will receive the potassium OXALATE 5%
  * Gingival dam will be performed using a fluid resin (Top Dam, FGM, Brazil) desensitivity gel application on vestibular surface, for 10 minutes.
  * A 35% hydrogen peroxide based bleaching agent will be mixed and applied on the vestibular surface of teeth, remaining for 40 minutes.
  Arms: Intervention: Potassium Oxalate 5% gel

SUMMARY:
Objectives: This study will determine the effectiveness of the use of desensitivity gels prior in office bleaching on risk and intensity of tooth sensitivity caused by in-office bleaching using 35% hydrogen peroxide. Materials and Methods: Fourty seven patients will be selected for this triple-blind, randomized, cross-over, placebo-controlled clinical trial. 10 minutes prior to bleaching procedure, patients will receive the the potassium nitrate 2% and potassium oxalate 5% desensitivity gel application on vestibular surface. The whitening treatment with 35% hydrogen peroxide will be carried out in two sessions with a 7-day interval. Tooth sensitivity will be assessed before, during and 24 hours after the procedure using analog visual and verbal scales. Color alteration will be assessed by a bleach guide scale and Vita Easy shade spectrophotometer 7 days after each session. Relative risk to sensitivity will be calculated and adjusted by session; while comparison of overall risk will performed by McNemar's test. Data on the sensitivity level for both scales and color shade will be subjected to the Friedman, Wilcoxon and Mann-Whitney tests, respectively (α = 0.05).

DETAILED DESCRIPTION:
Methods & Materials:

This clinical trial was approved by the Scientific Review Committee and by the Committee for the Protection of Human Subjects of the local university (CAAE 60259316.2.0000.5546).

Trial design:

This study will be a randomized, triple-blinded, placebo-controlled clinical trial, and split mouth study design.

The patients included will be submitted to two in-office bleaching sessions receiving the potassium nitrate 2% and postassium oxalate 5% desensitivity gel application on vestibular surface, for 10 minutes. A delay of 1 week between the sessions will be established. The study will be conducted at the clinic of the School of Dentistry of the local university from November 2016 to October 2017.

Participants:

Patients included in this clinical trial will be at least 18 years old with good oral health. Patients with any of the six upper anterior teeth with caries, restoration, severe discoloration (e.g., stains caused by tetracycline), enamel hypoplasia, gingival recession, dentin exposure, pulpitis, or endodontics will be excluded. Participants submitted to previous bleaching procedures, presenting prior tooth sensitivity, known allergy to any component of medication used in the study, pregnant or breastfeeding will be also excluded. Only patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (Vita Bleachguide 3D-Master scale, Vita-Zahnfabrik, Bad Sackingen, Germany) or darker will be included.

Sample Size Calculation:

The sample calculation will be based on the primary binary outcome (sensitivity risk 24 hours after the procedure) for superiority trial. Power of the test will be set at 80%, considering a type I error of 0.05; risk to tooth sensitivity of 63% (potassium nitrate) and 35% (potassium oxalate), while a reduction around 55% with the treatment will be expected. The calculation resulted in fourty seven patients.

Randomization:

A randomized list will be computer-generated by a person not involved in intervention or evaluation. The participants were defined as blocks in the randomization process, where the sequence of treatment (placebo or etodolac) will be randomly set for each block by using computer-generated tables (www.sealedenvelope.com). The sequence will be inserted into sealed envelopes numbered from 1 to 47 that were opened by the operator only at the moment of the intervention. The patients were numbered according to the sequence of enrollment. Neither the participant nor the operator knew the group allocation determining blinding to the protocol.

Baseline evaluation:

Prior to bleaching procedure, the teeth will be cleaned using rubber cups associated to pumice and water. The shades of six upper anterior teeth will be assessed on a baseline using the bleach guide scale and for CIE L*a*b* measurement, ΔE will be calculated by the following equation: ∆E= [(∆L)2 + (∆a)2 + (∆b)2]1/2, while ∆L = L1 - L0; ∆a = a1 - a0; e ∆b = b1 - b0.

Intervention:

Prior to each bleaching session, the patients will receive the potassium nitrate 2% (active comparator) on one half (anterior superior teeth) and potassium oxalate 5% desensitivity gel on the other half (anterior superior teeth) application on vestibular surface, for 10 minutes.

Neither the operators responsible for intervention and evaluation nor the patients knew the content which treatment will be done.

A light-cured resin dam will be applied (Top Dam, FGM, Joinville, SC, Brazil) on the gingival tissue corresponding to the teeth to be bleached. A 35% hydrogen peroxide based bleaching agent (Whiteness HP MAxx Intermixx, FGM, Joinville, SC, Brazil) will be mixed and applied on the vestibular surface of teeth, remaining for 40 minutes. After this time, the bleaching agent will be removed. A second session will be carried out after 1 week following the same procedures.

Evaluations:

The tooth sensitivity reported by patients will be assessed using a visual analog scale (VAS) and verbal rating scale (VRS). The VAS consisted of a scale 10 cm in length ranging from green (absence of pain) to red (unsupportable pain). The patient set his or her level of sensitivity by pointing to the color corresponding to this level, while the distance from this point to the green border will be recorded. For VRS, the patient reported his or her level of sensitivity based on scores: 0 = none, 1 = light, 2 = moderate, 3 = considerable and 4 = severe. The tooth sensitivity will be assessed during the bleaching, immediately after bleaching agent removal and after 24 hours. For this last assessment, only the VRS will be used. Tooth sensitivity will be measure: baseline, at 40 minutes during the bleaching procedure, after the bleaching procedure and 24 hours after. One week after each session the tooth color will be evaluated again using the same procedure described previously.

Statistical Analysis:

The demographic data from patients will be analyzed to determine age, gender, and anxiety level for each allocation sequence. Comparisons between the allocation sequences will be performed by the Mann-Whitney test (age) and Fisher's exact (gender) and chi-square (anxiety level) tests.

Based on presence of any tooth sensitivity (scores different from 0 for VRS), the absolute risk, odds ratio and relative risk will be calculated regarding the treatments for each moment of evaluation/session of bleaching, as well as its confidence intervals (95%). For each moment, differences on presence/absence ratios will be analyzed by Fisher's exact test. For the overall risk related to each treatment, the odds ratio will be adjusted to independent variable "session of bleaching" using the Mantel-Haenszel statistic. The homogeneity of odds ratios will be analyzed by the Breslow-Day and Tarone's tests. Following, the odds ratio estimated will be converted to relative risk and the overall presence/absence ratios will be analyzed by the McNemar's test, considering the study design (cross-over).

For VRS, the data from scores observed in each time of evaluation/session of bleaching will be submitted to the Mann-Whitney rank sum test. Despite the measurement of tooth sensitivity using VAS giving a continuous outcome, data assessed with this scale did not show a normal distribution (Shapiro-Wilk's test). Thus, data from VAS will be also analyzed by the Mann-Whitney rank sum test, while one test per time of evaluation will be carried out.

For color evaluation, comparisons between the sequences of treatment will be performed using the Mann-Whitney rank sum test. The Friedman test followed by Dunn's post hoc test will be used to analyze the difference between the moments of evaluation for each sequence of treatment. All statistical analyses will be performed adjusting the initial significance level (α = 0.05) by Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this clinical trial will be at least 18 years old with good oral health;
* Patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (Vita Bleachguide 3D-Master scale, Vita-Zahnfabrik, Bad Sackingen, Germany) or darker will be included.

Exclusion Criteria:

* Patients with any of the six upper anterior teeth with caries;
* Restorations in anterior teeth'
* Patients with tooth severe discoloration (e.g., stains caused by tetracycline);
* Presence of enamel hypoplasia;
* Presence of gingival recession or dentin exposure;
* Presence of tooth pulpitis or endodontics;
* Participants submitted to previous bleaching procedures;
* Patients with prior tooth sensitivity;
* Patients with known allergy to any component of medication used in the study;
* Pregnant or breastfeeding will also be also excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Risk to the tooth sensitivity | During the bleaching treatment.
  The tooth sensitivity will be assessed using a Visual analogue (VAS) and verbal scales. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper. The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Level of tooth sensitivity | During the Bleaching procedure
  The tooth sensitivity will be assessed using a Visual analogue (VAS) and verbal scales. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper.The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.
Risk after tooth sensitivity- after the procedure | 24 hours after the Bleaching procedure
  The tooth sensitivity will be assessed using a Visual analogue (VAS) and verbal scales. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper.The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated
Level of tooth sensitivity - after the procedure | 24 hours after the Bleaching procedure
  The tooth sensitivity will be assessed using a Visual analogue (VAS) and verbal scales. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper.The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.
Bleaching Effectiveness | Before the bleaching procedures and 7 days after this
  The color evaluation will be performed using CIE L*a*b* color system, classical Vita guide and Vita bleachguide. For the CIE L*a*b* and classical vita guide, the shade will be determined using a spectrophotometer (Easy Shade Compact, Vita-Zahnfabrik, Bad Säckinge, Germany). The spectrophotometer also will inform the shade in classical Vita guide.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Pardo S Nahsan, PhD, Principal Investigator — Universidade Federal de Sergipe
Locations (1):
- Flavia Pardo Salata Nahsan, Aracaju, Sergipe, Brazil

IPD SHARING:
Plan to Share IPD: No